CLINICAL TRIAL: NCT02894034
Title: Is the Measured Diameter of the Optic Nerve Sheath by Cerebral Scan in Patients With Early Phase Meningeal Hemorrhage Due to a Ruptured Aneurysm a Prognostic 6-month Mortality Factor?
Brief Title: Is the Measured Diameter of the Optic Nerve Sheath by Cerebral Scan in Patients With Early-phase Meningeal Hemorrhage, Due to a Ruptured Aneurysm, a Prognostic 6-month Mortality Factor ?
Acronym: GAINE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2013_843_0009
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Subarachnoid Hemorrhage
Keywords: optic nerve sheath; meningeal hemorrhage; early phase; prognostic
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Sub Arachnoid Hemorrhage (SAH) is a public health concern because of its high incidence (7/100 000 inhab.), its mortality rate (25%), and its morbidity rate (50%).

DETAILED DESCRIPTION:
Sub Arachnoid Hemorrhage (SAH) is a public health concern because of its high incidence (7/100 000 inhab.), its mortality rate (25%), and its morbidity rate (50%).

Prognostic tools are indispensable in guiding and optimizing the care of these patients.

Some diagnostic factors have been identified (e.g. age, comorbidities, ACSOS , GCS, ICP, occurrence of complications) as well as some classification schemes used for grading seriousness of the disease (Hunt and Hess, World Federation of NeuroSurgery).

A tool that is simple, reliable, reproducible, non costly, non invasive, and simple to perform (including remote methods and without changing planned patient care) would be ideal.

The measurement of the Optic Nerve Sheath Diameter (ONSD,) correlated by MRI and ultrasound in previous studies, with intra-cranial pressure (ICP: a fundamental prognostic factor for SAH) could be one of these tools.

This measurement, previously demonstrated using ultrasound, could be carried out at the time of the patient's initial cerebral scan.

In practice, at admission each patient undergoes a cerebral CT scan much more often than an ultrasound (faster, less costly, less technical training required).

Two preliminary studies seem to suggest that this measurement of ONSD on CTc is a predictive factor for morbi-morbidity in patients having serious traumatic skull fractures.The measurement is reliable, reproducible, non invasive, and non costly, with good sensitivity and specificity.

Proving that it is also applicable to SAH could be particularly useful.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Patient admitted to the Neurosurgical Urgent Care Unit for SAH following a ruptured aneurysm
* Patients or one of their loved ones providing written informed consent
* Patients with healthcare coverage

Exclusion Criteria:

* Unavailability of a CTc in the initial phase (within the first 12 hours) or absence of 1-mm slices from the scan
* Trauma to the optic globe or optic nerve pathology
* Preexisting anomalies of ICP or history of neurosurgical cerebral pathologies
* SAH of non aneurysm origin (e.g. arterio-venous malformation (AVM), tumor, trauma, sepsis)
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to the Neurosurgical Urgent Care Unit for SAH following a ruputred aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2013-08-19 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
patient survival | month 6
  patient survival

CONTACTS AND LOCATIONS:
Overall Officials: Patrick JEANJEAN, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France